CLINICAL TRIAL: NCT03421002
Title: Determination of Plasmatic and CSF Levels of High Doses of Micafungin in Neonates Suffering From Systemic Candidiasis and/or Candida Meningitis
Brief Title: Determination of Levels of Micafungin in Neonates Suffering From Systemic Candidiasis and/or Candida Meningitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: IRCCS, Ospedale Pediatrico Bambino Gesu (Unknown)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9463-CL-6001; 2014-003087-20 (EudraCT Number); 800_OPBG_2014 (Other: Ospedale Pediatrico Bambino Gesu Clinical & Research Center)
Record Dates: First submitted 2018-01-09; First posted 2018-02-05 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Candidiasis, Systemic; Candida Meningitis
Keywords: candida meningitis; Mycamine; candidiasis, systemic; micafungin
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Micafungin (Experimental): Participants will receive micafungin 8 mg/kg per day via intravenous infusion for approximately 1 hour. Micafungin will be administered for a minimum of 14 days until 1 of the following conditions applied: •Negative results (absence of Candida growth) from at least 2 consecutive blood cultures and/or resolution of clinical and laboratory symptoms and reduction of mannan antigen blood level (< 125 pg/mL) are obtained. •In case of meningitis, hydrocephalus and external ventricular derivation, negative results (absence of Candida growth) from at least 2 consecutive cerebral spinal fluid (CSF) cultures associated with resolution of clinical and laboratory symptoms. •Interruption (including addition or switch to another antifungal agent or dosage change of micafungin) due to demonstration of therapy failure.
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — Participants will receive micafungin 8 mg/kg per day via intravenous infusion for approximately 1 hour.
  Other Names: Mycamine

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetic profile of micafungin administered to neonates suffering from systemic candidiasis. This study will also evaluate the proportion of success and of failure of the therapy with micafungin among treated neonates and will identify a conversion factor to relate plasma levels of micafungin into capillary and venous blood measured through blood samples from the heel and from a peripheral vein, collected simultaneously. Safety of micafungin in neonates will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Infection by systemic candidiasis Systemic candidiasis is diagnosed in case of worsening of clinical conditions while on therapy with antibiotics, in case of isolation of candida from at least one sample collected from a normally sterile site (Blood, CSF, Urine, Peritoneal Fluid) and/or from at least two non contiguous sites (tracheal aspirate, gastric aspirate, faeces) and/or positivity to candida through polymerase chain reaction (PCR)(Septifast test), associated with at least one clinical symptom (fever or hypothermia, mottled skin, feeding difficulties, muscular hypotonia or hypertonia, apnoea crisis, bradycardia, tachycardia, hypotension, dyspnea, polypnea, desaturation) and one laboratory symptom (white blood cell [WBC] ≤5000/mm3 or WBC ≥20.000/mm3, immature to total neutrophil ratio [I/T ratio] >2, Platelet count ≤100.000/mm3, C-reactive Protein >0,5 mg/dL, Standard Base Excess >-7 mmol/L, CSF pleocytosis-cells ≥ 6) and/or positivity to test Enzyme Linked Immuno-Sorbent Assay (ELISA) for the mannan antigen (≥125 pg/ml).
* Neonates affected by candida meningitis and/or hydrocephalus due to candida infection and/or bearing external ventricular derivation, until enrollment of at least 4 subjects with this characteristics.
* Parents of neonates, or legal representative, able to consent and comply with protocol requirements.
* Survival expectation not inferior to 3 days.

Exclusion Criteria:

* Acute hepatopathy (ammonium > 200 µg/dL) or chronic hepatopathy.
* Known allergy or hypersensitivity to echinocandins or any of the excipients present in the formulation of the investigational product.

Ages: 1 Day to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2015-05-30 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Concentration of Micafungin in Blood | Predose and after 1, 3, and 8 hours post-dose on one of treatment days from Day 3 to Day 10
  Concentration will be determined from the pharmacokinetic (PK) blood samples collected via capillary micro-method (draws from the heel).
Concentration of Micafungin in Cerebral Spinal Fluid (CSF) | Predose and after 1, 3, and 8 hours post-dose on one of treatment days from Day 3 to Day 10
  Concentration will be determined from the from the CSF samples collected.

SECONDARY OUTCOMES:
Percentage of Participants with a Response at End of Treatment (EOT) - Success of Therapy (SOT) | Up to day 14
  For systemic candidiasis (SC) participants, SOT will be determined by survival associated with negative Candida test results of 2 consecutive blood cultures, completed at start of treatment, or resolution of clinical & laboratory symptoms together with reduction of mannan antigen blood level (MABL) (<125 pg/ml). For Candida meningitis (CM), SOT will be determined by survival associated with negative Candida test results of at least 2 consecutive CSF cultures, completed at start of treatment and resolution of clinical and lab symptoms. For hydrocephalus due to Candida infection (CI) and/or external ventricular derivation (EVD), SOT will be determined by survival associated with negative Candida test results of at least 2 consecutive CSF cultures, completed at start of treatment.
Percentage of Participants with A Response at EOT - Failure of Therapy (FOT) | Up to day 14
  For SC participants, FOT will be determined by death due to Candida sepsis, by confirmation of persistence of positive Candida test results from 1 blood culture completed by need to add/switch to another antifungal agent (AA) and/or change of micafungin dose for resolution of infection at any time or by the persistence of Candida colonization in different indicated sites associated with persistence of clinical and lab symptoms and with high (MABL) (≥ 125 pg/ml). For CM, FOT will be determined by death due to CM, by persistence of CI from confirmation of positive CSF culture or by need to add/switch to another AA or dose change of micafungin for resolution of CI at any time. For hydrocephalus due to CI and/or EVD, FOT will be determined by death due to CI, by need to add/switch to another AA or dose change of micafungin for resolution of CI at any time or by persistence of CI from confirmation of positive CSF culture.
Number of Participants with Adverse Events (AEs) | From the first dose of study drug administration up 72 hours after the last dose, up to 17 days
  An adverse event (AE) will be defined as any untoward medical occurrence in a participant administered a study drug or who will undergo study procedures which may not necessarily have a causal relationship with this treatment. This includes abnormal laboratory tests, vital signs, electrocardiogram data or physical examinations that are defined as AEs if the abnormality will induce clinical signs or symptoms, require active intervention, interruption or discontinuation of study drug or may be clinically significant in the investigator's opinion. The following standard with 3 grades will be used to measure the severity of AEs, including abnormal clinical laboratory values: ● Mild: No disruption of normal daily activities ● Moderate: Affected normal daily activities ● Severe: Inability to perform daily activities. A treatment-emergent adverse event (TEAE) will be defined as an AE observed after starting administration of the test drug/comparative drug.
Comparison of Capillary and Venous Plasma Concentrations of Micafungin | Predose and after 1, 3, and 8 hours post-dose on one of treatment days from Day 3 to Day 10
  Micafungin concentrations will be determined from the PK blood samples collected via both capillary micro-method (draws from the heel) and venous methods.

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (2):
- Italy (2):
  - Site IT39001, Rome
  - Site IT39002, Rome

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Auriti C, Goffredo BM, Ronchetti MP, Piersigilli F, Cairoli S, Bersani I, Dotta A, Bagolan P, Pai MP. High-Dose Micafungin in Neonates and Young Infants with Invasive Candidiasis: Results of a Phase 2 Study. Antimicrob Agents Chemother. 2021 Mar 18;65(4):e02494-20. doi: 10.1128/AAC.02494-20. Print 2021 Mar 18. PMID 33558294
- See also: Link to Results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=312